CLINICAL TRIAL: NCT03253094
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Double-Dummy, Active-Controlled, Dose-Finding Study to Compare the Safety and Efficacy of Oral Ibrexafungerp (SCY-078) vs. Oral Fluconazole in Subjects With Acute Vulvovaginal Candidiasis
Brief Title: Dose-Finding Study of Oral Ibrexafungep (SCY-078) vs. Oral Fluconazole in Subjects With Acute Vulvovaginal Candidiasis
Acronym: DOVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCY-078-204
Record Dates: First submitted 2017-07-14; First posted 2017-08-17 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Candida Vulvovaginitis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole; ibrexafungerp

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, double-dummy, active-controlled, dose-finding
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Fluconazole (Active Comparator): 150 mg/day for 1 day
  Interventions: Drug: Fluconazole
- Ibrexafungerp 750mg (Experimental): 750mg QD for 1 day only
  Interventions: Drug: SCY-078
- Ibrexafungerp 300mg (Experimental): 300mg BID for 1 day only
  Interventions: Drug: SCY-078
- Ibrexafungerp 450mg (Experimental): 450mg BID for 1 day only
  Interventions: Drug: SCY-078
- Ibrexafungerp 150mg (Experimental): 150mg BID for 3 days
  Interventions: Drug: SCY-078
- Ibrexafungerp 300mg D1-D3 (Experimental): 300mg BID for 3 days
  Interventions: Drug: SCY-078

INTERVENTIONS:
Drug: Fluconazole — Oral Antifungal comparator
  Other Names: Diflucan, Azole antifungal
  Arms: Fluconazole
Drug: SCY-078 — Investigational Antifungal
  Other Names: Ibrexafungerp
  Arms: Ibrexafungerp 150mg; Ibrexafungerp 300mg; Ibrexafungerp 300mg D1-D3; Ibrexafungerp 450mg; Ibrexafungerp 750mg

SUMMARY:
This is a multicenter, randomized, double-blind, double-dummy, active-controlled, dose-finding study to compare the efficacy, safety and tolerability of oral SCY-078 versus oral fluconazole in adult female subjects 18 years and older with moderate to severe Acute Vulvovaginal Candidiasis (AVVC). Approximately 180 eligible subjects (30 subjects per treatment group) will be enrolled and randomized into the study.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, double-dummy, active-controlled, dose-ranging study of female subjects with moderate to severe Acute Vulvovaginal Candidiasis. Subjects will be randomized to either the investigational arm (SCY-078) with 5 different dose regiments ranging from 1 to 3 days of treatment or to the active-control arm (fluconazole) for 1 day of treatment. After randomization subjects may be seen on study Day 3 (on site visit for PK subjects) , Day 10 (±2,) and Day 25 (+4).

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject is a female of at least 18 years of age
2. Subject has a diagnosis of symptomatic AVVC at baseline including a positive microscopic examination with 10% KOH in a vaginal sample revealing yeast forms (hyphae/pseudohyphae) or budding yeasts, and vaginal pH (≤4.5)

Key Exclusion Criteria:

1. Subject has any vaginal condition other than AVVC that may interfere with the diagnosis or evaluation of response to therapy, such as suspected or confirmed concurrent causes of vulvovaginitis and/or cervicitis (mixed infection)
2. Need for systemic and/or topical (vaginal) antifungal treatment, including prescription or over-the-counter products during the study and treatment for VVC 28 days prior to randomization
3. Subject is actively menstruating at the time of the Baseline visit.
4. Subject has uncontrolled diabetes mellitus.
5. Subject has a vaginal sample with pH >4.5.
6. Subject has a history of or an active cervical/vaginal cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 186 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Angulo, MD, Study Director — Scynexis, Inc.
Locations (25):
- United States (25):
  - UAB Personal Health Clinic, Birmingham, Alabama
  - Precision Trials AZ, LLC, Phoenix, Arizona
  - Women's Health Care Research Corp., San Diego, California
  - Gulf Coast Research Group, LLC, Brandon, Florida
  - Altus Research, Inc., Lake Worth, Florida
  - OB-GYN Associates of Mid-Florida P.A., Leesburg, Florida
  - New Age Medical Research Corp., Miami, Florida
  - Visionary Investigators Network, South Miami, Florida
  - Atlanta North Gynecology, P.C., Roswell, Georgia
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Clinical Trials Management, LLC, Covington, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Women Under Study, LLC, New Orleans, Louisiana
  - Tolan Park Medical Building, Detroit, Michigan
  - Consultants in Women's Healthcare, Inc., St Louis, Missouri
  - Lawrence OB/GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - Women's Health Research Center, Plainsboro, New Jersey
  - Unified Women's Clinical Research - Central Carolina, Greensboro, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Drexel University, Philadelphia, Pennsylvania
  - Medical Research South, LLC, Charleston, South Carolina
  - WR-Medical Research Center of Memphis, LLC, Memphis, Tennessee
  - Tmc Life Research, Inc., Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Seattle Women's Health, Research, Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nyirjesy P, Schwebke JR, Angulo DA, Harriott IA, Azie NE, Sobel JD. Phase 2 Randomized Study of Oral Ibrexafungerp Versus Fluconazole in Vulvovaginal Candidiasis. Clin Infect Dis. 2022 Jul 6;74(12):2129-2135. doi: 10.1093/cid/ciab841. PMID 34555149

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrexafungerp 750-mg: 750 mg QD for 1 day only
- Ibrexafungerp 300-mg: 300 mg BID for 1 day only
- Ibrexafungerp 450-mg: 450 mg BID for 1 day only
- Ibrexafungerp 150-mg: 150 mg BID for 3 days
- Ibrexafungerp 300-mg (3 Days): 300 mg BID for 3 days
- Fluconazole: 150 mg QD for 1 day
Period: Overall Study
Arm/Group | Ibrexafungerp 750-mg | Ibrexafungerp 300-mg | Ibrexafungerp 450-mg | Ibrexafungerp 150-mg | Ibrexafungerp 300-mg (3 Days) | Fluconazole
Started | 32 | 30 | 28 | 32 | 32 | 32
Subjects Discontinued | 4 | 3 | 6 | 4 | 5 | 4
Completed | 28 | 27 | 22 | 28 | 27 | 28
Not Completed | 4 | 3 | 6 | 4 | 5 | 4
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 3 | 0
Not completed — Other | 0 | 1 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrexafungerp 750-mg | Ibrexafungerp 300-mg | Ibrexafungerp 450-mg | Ibrexafungerp 150-mg | Ibrexafungerp 300-mg (3 Days) | Fluconazole | Total
Number analyzed (Participants) | 32 | 30 | 28 | 32 | 32 | 32 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (12.3) | 34.4 (11.3) | 34.5 (9.8) | 33.3 (10.5) | 32.0 (8.5) | 33.8 (10.1) | 33.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 28 | 32 | 32 | 32 | 186
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 8 | 11 | 7 | 11 | 56
  Not Hispanic or Latino | 22 | 21 | 20 | 21 | 25 | 21 | 130
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 10 | 12 | 13 | 15 | 13 | 72
  White | 22 | 20 | 14 | 18 | 16 | 19 | 109
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 28 | 32 | 32 | 32 | 186

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure (Complete Resolution of Signs and Symptoms)
Description: Measured by the percentage of subjects with clinical cure (complete resolution of signs and symptoms) at the test-of-cure (TOC) visit
Time Frame: 8-12 days
Population: mITT
Measure: Count of Participants; unit: Participants
Groups:
- Ibrexafungerp 750-mg: 750 mg QD D1 only
- Ibrexafungerp 300-mg: 300 mg BID D1 only
- Ibrexafungerp 450-mg: 450 mg BID D1 only
- Ibrexafungerp 150-mg: 150 mg BID D1 to D3
- Ibrexafungerp 300-mg D1 to D3: 300 mg BID D1 to D3
- Fluconazole: 150 mg QD D1 only
Arm/Group | Ibrexafungerp 750-mg | Ibrexafungerp 300-mg | Ibrexafungerp 450-mg | Ibrexafungerp 150-mg | Ibrexafungerp 300-mg D1 to D3 | Fluconazole
Number analyzed (Participants) | 26 | 27 | 21 | 29 | 26 | 24
Participants
  Clinical cure | 9 | 14 | 13 | 14 | 15 | 14
  Clinical failure | 17 | 13 | 8 | 15 | 11 | 10

2. Secondary Outcome: Co-occurrence of Clinical and Mycological Cure
Description: The percentage of subjects with both clinical cure and mycological eradication (negative fungal culture) the Test-of cure.
Time Frame: 29 days
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 750-mg | Ibrexafungerp 300-mg | Ibrexafungerp 450-mg | Ibrexafungerp 150-mg | Ibrexafungerp 300-mg D1 to D3 | Fluconazole
Number analyzed (Participants) | 26 | 27 | 21 | 29 | 26 | 24
Participants
  Clinical cure and Mycological Eradication | 4 | 10 | 11 | 8 | 13 | 10
  Clinical failure and/or mycological persistence | 22 | 17 | 10 | 21 | 13 | 14

3. Other Pre Specified Outcome: Incidence of Treatment Emergent Adverse Events
Description: The number of subjects with treatment related adverse events
Time Frame: up to 29 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 750-mg | Ibrexafungerp 300-mg | Ibrexafungerp 450-mg | Ibrexafungerp 150-mg | Ibrexafungerp 300-mg D1 to D3 | Fluconazole
Number analyzed (Participants) | 32 | 30 | 28 | 31 | 32 | 32
Participants
  Treatment related Treatment-emergent adverse event | 20 | 14 | 16 | 12 | 15 | 8
  No Treatment related Treatment-emergent adverse event | 12 | 16 | 12 | 19 | 17 | 24

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | Ibrexafungerp 750-mg | Ibrexafungerp 300-mg | Ibrexafungerp 450-mg | Ibrexafungerp 150-mg | Ibrexafungerp 300-mg D1 to D3 | Fluconazole
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30 | 0/28 | 0/31 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30 | 0/28 | 0/31 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 21/32 | 13/30 | 15/28 | 15/31 | 18/32 | 10/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp 750-mg (N=32) | Ibrexafungerp 300-mg (N=30) | Ibrexafungerp 450-mg (N=28) | Ibrexafungerp 150-mg (N=31) | Ibrexafungerp 300-mg D1 to D3 (N=32) | Fluconazole (N=32)
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 2 | 3 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 15 | 5 | 6 | 4 | 13 | 1
Nausea (Gastrointestinal disorders) | 8 | 3 | 8 | 6 | 6 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 4 | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 0 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 2 | 3 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 3 | 9 | 4 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 2 | 2 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03253094/Prot_001.pdf
  • Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT03253094/SAP_002.pdf